CLINICAL TRIAL: NCT02886234
Title: Mindfulness Training to Improve ART Adherence and Reduce Risk Behavior Among Persons Living With HIV
Brief Title: Health Improvement Project - Providence
Acronym: HIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Michael P. Carey, Professor and Director, Centers for Preventive and Behavioral Medicine, The Miriam Hospital, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34AT008930 (NIH); R34AT008930 (NIH)
Record Dates: First submitted 2016-08-18; First posted 2016-09-01 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: HIV
Keywords: HIV; Mindfulness; Adherence behaviors; Stress; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness training (MT) (Experimental): Eight, 30-minute phone delivered MT sessions once a week for 8 weeks
  Interventions: Behavioral: Mindfulness Training (MT)
- Health Coaching (HC) (Active Comparator): Eight, 30-minute phone delivered HC sessions once a week for 8 weeks
  Interventions: Behavioral: Health Coaching (HC)

INTERVENTIONS:
Behavioral: Mindfulness Training (MT) — Participants assigned to the MT condition will receive a phone-delivered 30-minute mindfulness training once a week for 8 weeks. ). In addition to the weekly training session, participants will be instructed to practice mindfulness techniques for 15 minutes daily using a standardized audio recording to guide the participant through the techniques learned with the instructor.
  Arms: Mindfulness training (MT)
Behavioral: Health Coaching (HC) — The HC condition will consist of educational modules designed to control for the contact time and attention received in the MT condition. To match the time MT participants will spend doing mindfulness exercises at home, HC participants will be assigned a 15-minute daily activity that is aligned with the HC topics
  Arms: Health Coaching (HC)

SUMMARY:
This study will investigate whether phone-delivered mindfulness training is feasible and acceptable for persons living with HIV and whether it may help them improve adherence to medications and reduce risky sexual behaviors.

DETAILED DESCRIPTION:
Two-thirds of people living with HIV show sub-optimal adherence to antiretroviral therapy (ART) and one-third engages in risky sex. Both non-adherence and risky sex have been associated with emotional distress and impulsivity. In this trial, the investigators will examine the utility of phone-delivered mindfulness training (MT) for people living with HIV. The primary outcomes comprise feasibility and acceptability of phone-delivery; secondary outcomes are estimates of efficacy of MT on adherence to ART and safer sexual practices as well as on their hypothesized antecedents.

Fifty participants will be enrolled in this parallel-group randomized clinical trial (RCT). Outpatients recruited from an HIV treatment clinic will be randomized (1:1 ratio) to either MT or to health coaching intervention; both interventions will be administered during 8 weekly phone calls. ART adherence (self-reported measure and unannounced phone pill counts), sexual behavior (self-reports and biomarkers), mindfulness, depression, stress, and impulsivity will be measured at baseline, post-intervention, and 3 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Sub-optimal adherence to ART (Less than "always" taking ART medication and/or viral load > 20 copies/mL);
* Psychological distress (PHQ-4 score ≥ 2);
* Recent risky sexual behavior (any unprotected sex OR > 1 sexual partner over the past 6 months)
* Access to a telephone or cell phone

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* Cognitive impairment
* Non-English speaking
* Low literacy (i.e., reporting they "often" or "always" need someone to read instructions, pamphlets, or other written material from a doctor or pharmacy to them
* Enrolled in another behavioral trials
* Prior formal mindfulness training or have practiced of mindfulness or related mind-body techniques in the previous year
* Severe hearing impairment not allowing phone delivery
* Suicidal ideation
* Planning to move out of the area within the study period
* Clinic provider advising against recruitment in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MIchael P Carey, PhD, Principal Investigator — Centers for Behavioral and Preventive Medicine, The Miriam Hospital; Elena Salmoirago-Blotcher, MD, PhD, Principal Investigator — Centers for Behavioral and Preventive Medicine, The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to being randomized, patients had to complete all baseline activities, which included two months of counting to establish a baseline adherence measure. During this interval, 6 patients withdrew from the study. Thus, 44 patients were randomized (24 to health coaching arm, and 20 to the mindfulness training arm).
Period: Overall Study
Arm/Group | Mindfulness Training (MT) | Health Coaching (HC)
Started | 20 | 24
Completed | 20 | 22
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Training (MT) | Health Coaching (HC) | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (11.7) | 48.5 (11.0) | 47.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 7 | 11
  White | 10 | 8 | 18
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Intervention
Description: Feasibility - as indicated by the number of patients attending at least 50% of sessions
Time Frame: post-intervention, 9 to 10 weeks after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Training (MT) | Health Coaching (HC)
Number analyzed (Participants) | 20 | 22
Participants | 11 | 19

2. Secondary Outcome: Acceptability of the Intervention
Description: Number of patients reporting "very satisfied" or "mostly satisfied" with their intervention
Time Frame: post-intervention, 9 to 10 weeks after baseline
Population: 3 participants in the MT arm did not complete the acceptability rating at the post-intervention assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Training (MT) | Health Coaching (HC)
Number analyzed (Participants) | 17 | 22
Participants | 15 | 19

3. Secondary Outcome: Antiretroviral Medication Adherence
Description: Self-reported number of missed days of medication
Time Frame: Baseline; post-intervention, 9 to 10 weeks after baseline; follow-up, 21 to 22 weeks after baseline
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mindfulness Training (MT) | Health Coaching (HC)
Number analyzed (Participants) | 20 | 22
days
  Baseline | 4.20 (7.02) | 1.95 (3.15)
  Post-Intervention | 3.41 (6.57) | 1.64 (3.30)
  3-month Follow-up | 2.70 (3.53) | 1.45 (1.99)

4. Secondary Outcome: Self-reported Sexual Risk Behavior
Description: Self-reported risky sexual behavior as indicated by the percentage of episodes of condom protected sexual intercourse Higher values are better outcome
Time Frame: Baseline; post-intervention, 9 to 10 weeks after baseline; follow-up, 21 to 22 weeks after baseline
Measure: Mean (Standard Deviation); unit: percentage of sexual events condom used
Arm/Group | Mindfulness Training (MT) | Health Coaching (HC)
Number analyzed (Participants) | 20 | 22
percentage of sexual events condom used
  Baseline | 57 (44) | 32 (44)
  post-intervention | 100 (236) | 49 (71)
  3-month Follow-up | 71 (49) | 43 (48)

5. Secondary Outcome: Five Facet Mindfulness Questionnaire
Description: Five Facet of Mindfulness Questionnaire (15 items; short form) Construct = Mindfulness Minimum total scale score = 15 Maximum total scale score = 75 Scoring: sum across all 15 items Higher scores represent a better outcome
Time Frame: Baseline; post-intervention, 9 to 10 weeks after baseline; follow-up, 21 to 22 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT) | Health Coaching (HC)
Number analyzed (Participants) | 20 | 22
score on a scale
  Baseline | 47.70 (7.09) | 49.09 (8.09)
  Post-Intervention | 53.06 (10.32) | 52.73 (8.98)
  3-month Follow-up | 53.05 (7.49) | 52.18 (7.84)

6. Secondary Outcome: Perceived Stress Scale
Description: Perceived Stress Scale (4-item version) Construct = perceived stress Minimum total scale score = 0 Maximum total scale score = 16 Scoring: reverse score items 2 and 3, then sum across all 4 items Higher scores represent a worse outcome
Time Frame: Baseline; post-intervention, 9 to 10 weeks after baseline; follow-up, 21 to 22 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT) | Health Coaching (HC)
Number analyzed (Participants) | 20 | 22
score on a scale
  Baseline | 6.90 (4.09) | 5.86 (3.01)
  post-Intervention | 6.06 (3.58) | 5.64 (2.75)
  3-month Follow-up | 5.80 (3.71) | 5.73 (3.28)

7. Secondary Outcome: Barratt Impulsiveness Scale
Description: Barratt Impulsiveness Scale (short form, 8 items) Construct = Impulsivity Minimum total scale score = 8 Maximum total scale score = 32 Scoring: reverse score items 1, 4, 5, 6, and then sum across all 8 items Higher scores represent a worse outcome
Time Frame: Baseline; post-intervention, 9 to 10 weeks after baseline; follow-up, 21 to 22 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT) | Health Coaching (HC)
Number analyzed (Participants) | 20 | 22
score on a scale
  baseline | 18.15 (3.76) | 17.50 (4.36)
  post-intervention | 17.76 (4.31) | 15.68 (3.40)
  3-month Follow-up | 16.05 (4.07) | 16.50 (4.42)

8. Secondary Outcome: Patient Health Questionnaire
Description: Patient Health Questionnaire (9 item version) Construct measured = depression Minimum total scale score = 0 Maximum total scale score = 27 Scoring: sum across all 9 items Higher scores represent a worse outcome
Time Frame: Baseline; post-intervention, 9 to 10 weeks after baseline; follow-up, 21 to 22 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT) | Health Coaching (HC)
Number analyzed (Participants) | 20 | 22
score on a scale
  Baseline | 9.80 (6.58) | 8.55 (5.54)
  Post-Intervention | 8.82 (6.66) | 5.68 (4.82)
  3-month Follow-up | 6.90 (5.23) | 5.18 (3.72)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the trial, starting at baseline and continuing through the initial pill count phase of baseline (2 months), the intervention period (2 months), and during the 3-month follow-up period (3 months). Thus, adverse events were monitored for a total of 7 months.
Arm/Group | Mindfulness Training (MT) | Health Coaching (HC)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 0/20 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT02886234/Prot_SAP_000.pdf
  • Informed Consent Form (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT02886234/ICF_001.pdf